CLINICAL TRIAL: NCT05118178
Title: Prognostic Significance of the Atherosclerosis in the Coronary Arteries Assessed in Computed Tomography on the Cardiotoxicity Development After Oncological Treatment
Brief Title: Atherosclerosis in Chemotherapy-related Cardiotoxicity
Acronym: ANTEC
Status: Completed | Type: Observational
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Polish Cardiac Society (Other); Servier (Industry)
Responsible Party: Principal Investigator, Anna Borowiec, Principal Investigator, Maria Sklodowska-Curie National Research Institute of Oncology
Other Study IDs: 80/2021
Record Dates: First submitted 2021-10-26; First posted 2021-11-11 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Cardiotoxicity; Atherosclerosis
MeSH Terms: conditions — Cardiotoxicity; Atherosclerosis | interventions — Echocardiography; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: echocardiography, computed tomography — echocardiography - including GLS and MWI computed tomography - with calcium score index

SUMMARY:
Cardiological complications of oncological treatment, including the most serious of them cardiotoxicity and heart failure, constitute a significant and still unsolved clinical problem. A history of hypercholesterolaemia and coronary artery disease in cancer patients, is one of the risk factors for cardiotoxicity. In recent years, a protective effect of statin treatment on the development of heart failure in cancer patients has been observed. ANTEC (Atherosclerosis iN chemoTherapy-rElated Cardiotoxicity) is a prospective observational study aimed at assessing the impact of the advancement of atherosclerotic lesions in the coronary arteries assessed in computed tomography on the development of left ventricular systolic dysfunction in cancer patients at high risk of myocardial damage. A group of 80 patients diagnosed with cancer before starting high-dose anthracycline chemotherapy (doxorubicin ≥ 240 mg / m2 or epirubicin ≥ 600 mg / m2 body weight), without a history of heart failure and coronary artery disease, will be included in the study. The total follow-up of patients was planned for 12 months. The primary endpoint is time to onset of left ventricular systolic dysfunction as assessed by echocardiography. The secondary composite endpoints include all-cause death, cardiovascular death, myocardial infarction, and stroke. Additionally, the assessment will include: the severity of atherosclerotic changes in the coronary arteries and the calcification index in computed tomography, the percentage decrease in left ventricular ejection fraction, GLS (global longitudinal strain) in echocardiography, and changes in the concentration of biomarkers involved in inflammatory and atherosclerotic processes. This is the first study of this type, which we hope will contribute to a better understanding of the pathophysiology of cardiotoxicity development and to changing the standards of management of oncological patients and improving survival in this group of patients.

DETAILED DESCRIPTION:
Cardiological complications of oncological treatment, including the most serious: cardiotoxicity and heart failure, remains the most dangerous cardiological complication of oncological treatment and are still unsolved clinical problem. The fear of the toxic effects of anti-cancer drugs may lead to the modification or abandonment of oncological treatment, and consequently shorten the survival time of cancer patients.

A history of hypercholesterolaemia and coronary artery disease in cancer patients, is one of the risk factors for cardiotoxicity. In recent years, a protective effect of statin treatment on the development of heart failure in cancer patients has been observed. ANTEC (Atherosclerosis iN chemoTherapy-rElated Cardiotoxicity) is a prospective observational study aimed at assessing the impact of the advancement of atherosclerotic lesions in the coronary arteries assessed in computed tomography on the development of left ventricular systolic dysfunction in cancer patients at high risk of myocardial damage. A group of 80 patients diagnosed with cancer before starting high-dose anthracycline chemotherapy (doxorubicin ≥ 240 mg / m2 or epirubicin ≥ 600 mg / m2 body weight), without a history of heart failure and coronary artery disease, will be included in the study. The total follow-up of patients was planned for 12 months. The primary endpoint is time to onset of left ventricular systolic dysfunction as assessed by echocardiography. The secondary composite endpoints include all-cause death, cardiovascular death, myocardial infarction, and stroke. Additionally, the assessment will include: the severity of atherosclerotic changes in the coronary arteries and the calcification index in computed tomography, the percentage decrease in left ventricular ejection fraction, GLS (global longitudinal strain) in echocardiography, and changes in the concentration of biomarkers involved in inflammatory and atherosclerotic processes. This is the first study of this type, which we hope will contribute to a better understanding of the pathophysiology of cardiotoxicity development and to changing the standards of management of oncological patients and improving survival in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.
2. Age ≥18 years at the time of signing the informed consent.
3. Known neoplastic disease prior to the initiation of chemotherapy with a high dose of anthracyclines (doxorubicin ≥ 240 mg / m2 b.w. or epirubicin ≥ 600 mg / m2 b.w.)
4. No history of heart failure (left ventricular ejection fraction ≥ 50% as assessed by echocardiography).
5. No history of: coronary artery disease, stroke and lower limb atherosclerosis
6. At least moderate baseline cardiovascular toxicity risk according to Heart Failure Association-International Cardio-Oncology Society stratification

Exclusion Criteria:

1. History of heart failure
2. Left ventricle systolic dysfunction with LVEF <50%
3. Significant valve defect
4. Previous chemotherapy or radiation to the chest
5. Presence of any disease with a life expectancy <1 year in the opinion of the investigator.
6. Drug or alcohol abuse
7. Lack of possibility or contraindications for coronary tomography before starting chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients with diagnosed cancer, diagnosed and qualified for further systemic treatment at the National Institute of Oncology in Warsaw. Patients must give informed and voluntary consent to participate in the study and meet all the conditions for inclusion in the study
  The size of the study group was calculated at 80 people. The estimated group size is based on the Cochran-Armitage test for the existence of a trend for a variable on an ordinal scale. The one-sided test was taken into account (alternative hypothesis - increase in the incidence of cardiotoxicity with the severity of atherosclerotic lesions versus null hypothesis - no effect). Assumptions: power - 80%, level of statistical significance - 0.05, one-tailed test for the presence of a trend.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Patients with left ventricular systolic dysfunction | from date of randomization until the end of study, up to 12 months
  echocardiography

SECONDARY OUTCOMES:
Time to the secondary composite endpoint: all-cause death, cardiovascular death, myocardial infarction, and stroke | from date of randomization until the end of study, up to 12 months
  medical records

OTHER OUTCOMES:
The presence of atherosclerosis in the coronary arteries and the calcification index | from date of randomization until the end of study, up to 12 months
  computed tomography
Percentage decrease in left ventricular ejection fraction, GLS (global longitudinal strain) and MWI (myocardial work index) | from date of randomization until the end of study, up to 12 months
  echocardiography
Changes in the concentration of biomarkers involved in inflammatory and proatherosclerotic processes (IL-6, MPO i TNF-alfa). | from date of randomization until the end of study, up to 12 months
  blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borowiec A, Ozdowska P, Rosinska M, Jagiello-Gruszfeld A, Jasek S, Waniewska J, Kotowicz B, Kosela-Paterczyk H, Lampka E, Makowka A, Fuksiewicz M, Chojnacka M, Zebrowska A, Gepner K, Kapala A, Cieszanowski A, Nowecki Z, Walewski J. Prognostic value of coronary atherosclerosis and CAC score for the risk of chemotherapy-related cardiac dysfunction (CTRCD): The protocol of ANTEC study. PLoS One. 2023 Aug 17;18(8):e0288146. doi: 10.1371/journal.pone.0288146. eCollection 2023. PMID 37590267